CLINICAL TRIAL: NCT04234256
Title: Controlled, Randomized, Stretching Exercises for Improvement of Dynamic Balance
Brief Title: Female Football Players Stretching Training and Performance on the Dynamic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dragan Mijatović (Other)
Responsible Party: Sponsor-Investigator, Dragan Mijatović, Master of Physiotherapy, Postgraduate Study in Health Sciences, University of Mostar
Organization: University of Mostar (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Study 3
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Stretch
Keywords: Y Balance Test; Stretching; Dynamic balance
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static exercise (Experimental): The experimental group doing static exercises, three times with five repetitions for a period of three months lasting 15 to 20 minutes at the end of the training.
  Interventions: Other: Static stretching exercise
- Dynamic exercise (Experimental): This group doing dynamic exercises, three times with five repetitions for a period of three months lasting 15 to 20 minutes at the end of the training.
  Interventions: Other: Dynamic stretching exercise
- Control group (No Intervention): Control group doing not the stretching exercise

INTERVENTIONS:
Other: Static stretching exercise — Standing quadriceps stretch, Gastrocnemius stretch, Standing split, Adductor stretch, Half kneeling groin stretch, Hamstring stretch on the bench, Prayer squat, Seated adductor and hamstring stretch, Hurdle seat, Seated glute stretch, Lying glute stretch, Seated groin abduction, Soleus stretch, Half kneeling quad stretch, Split hamstring stretch
  Arms: Static exercise
Other: Dynamic stretching exercise — Downward dog to runner's lunge, Dynamic squat stretch, Crescent to hamstring stretch, Half kneeling hamstring stretch, Side to side lunge with reach, Standing calf and hamstring stretch, Hurdles, Side to side lunge with step, IT band stretch, Walking quad stretch, Swing the leg forward and back, Swing the leg cross, Knee pull, Standing quat stretch, Standing gluteus stretch
  Arms: Dynamic exercise

SUMMARY:
This research shows the effect of stretching exercises on dynamic balance. football players divided into 2 groups do different stretching exercises, dynamic and static. The control group does not do stretching exercises. The study should show which stretching exercises have a greater effect on the Y balance test than the dynamic balance test.

DETAILED DESCRIPTION:
Injury prevention in sports is very important, and a lot of investigative time and effort is spent in this realm. Many different tools have been created that are designed to pinpoint the athlete's predisposition to or risk for injuries. Also, health professionals and coaches should work with athletes to attempt to reduce the number of injuries as much as possible. The objective of the prevention process is not to eliminate injuries, but rather to reduce them and keep them at an acceptable level. Many authors have shown that interventions that include balance exercises are very efficient in injury risk reduction as well as performance improvement after an injury. Poor balance, altered motor control, or lack of neuromuscular control have all been described as predictors of injury risk in the lower limbs of athletes. The Y-Balance Test (YBT), a validated derivation of the Star Excursion Balance Test (SEBT), is a functional screening tool that can be reliably administered for a variety of purposes: to assess lower extremity stability, monitor rehabilitation progress, understand deficits after injury, and identify athletes at high risk for lower extremity injury. For these reasons, we have decided to research whether stretching exercises can improve the Y Balance Test. The research was conducted on football players in the first league of Bosnia and Hercegovina. Comparisons were made between static and dynamic stretching and their effects on Y Balance Test performance while no stretching exercises were performed in the control group. Stretching improves body posture, achieves good muscular and joint mobility, has a positive effect on preventing injury, and reduces muscle pain, also regular stretching improves body balance. The aim is to explore which stretching exercises will increase the results on the Y Balance Test and whether this will happen at all.

This study aimed to investigate the effects of stretching exercises on the Y-Balance Test (YBT, as a test for dynamic balance) performance and postural control in female football players.

ELIGIBILITY:
Inclusion Criteria:

* No musculoskeletal injury within 10 days of the start of the study,
* Age over 14 years (The Official Gazette of the Football Federation of the Federation of Bosnia and Herzegovina, the Women's Football League of the Federation of Bosnia and Herzegovina, article 15. states that female players who have reached the age of 14 and who have a specialist medical examination can play for the first team, a maximum of 5 player's on the field in the same game)
* Voluntary participation in the study.

Exclusion Criteria:

* Age below 14 years,
* Refusal to take the examination,
* Errors in keeping records of injuries by responsible persons,
* Lower legs injuries in the last 10 days,
* Vestibular disorders.

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
The leg length | 2 minutes
  The leg length was measured from the anterior superior iliac spine to the distal edge of the medial malleolus, in centimeter using a tape measure.
Y Balance Test | 15 minutes
  During the test, the football players place one foot on the stationary platform of the test set so that the tip of the foot does not exceed the starting line. The second foot, or the tip of the foot, will push the movable part of the platform down the measuring tube, which is marked by half-inch intervals. Any lifting of the standing leg to the heel, toes or loss of balance will be considered a mistake and the attempt will be repeated. Mobility will be tested through 3 trial and 3 valid measurements of the lower limbs in the anterior, posteromedial, and posterolateral directions. The arms should rest on the hips.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan mijatović, MPT, Principal Investigator — WFC Siroki Brijeg
Locations (1):
- ŽNK Široki Brijeg, Široki Brijeg, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonell AC, Romero JA, Soler LM. RELATIONSHIP BETWEEN THE Y BALANCE TEST SCORES AND SOFT TISSUE INJURY INCIDENCE IN A SOCCER TEAM. Int J Sports Phys Ther. 2015 Dec;10(7):955-66. PMID 26673848
- [Background] Butler RJ, Bullock G, Arnold T, Plisky P, Queen R. Competition-Level Differences on the Lower Quarter Y-Balance Test in Baseball Players. J Athl Train. 2016 Dec;51(12):997-1002. doi: 10.4085/1062-6050-51.12.09. Epub 2016 Nov 16. PMID 27849388
- [Background] Hooper TL, James CR, Brismee JM, Rogers TJ, Gilbert KK, Browne KL, Sizer PS. Dynamic balance as measured by the Y-Balance Test is reduced in individuals with low back pain: A cross-sectional comparative study. Phys Ther Sport. 2016 Nov;22:29-34. doi: 10.1016/j.ptsp.2016.04.006. Epub 2016 May 4. PMID 27579805
- [Background] Fuller CW, Ekstrand J, Junge A, Andersen TE, Bahr R, Dvorak J, Hagglund M, McCrory P, Meeuwisse WH. Consensus statement on injury definitions and data collection procedures in studies of football (soccer) injuries. Scand J Med Sci Sports. 2006 Apr;16(2):83-92. doi: 10.1111/j.1600-0838.2006.00528.x. PMID 16533346
- [Background] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Background] Kinzey SJ, Armstrong CW. The reliability of the star-excursion test in assessing dynamic balance. J Orthop Sports Phys Ther. 1998 May;27(5):356-60. doi: 10.2519/jospt.1998.27.5.356. PMID 9580895
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Zakaria AA, Kiningham RB, Sen A. Effects of Static and Dynamic Stretching on Injury Prevention in High School Soccer Athletes: A Randomized Trial. J Sport Rehabil. 2015 Aug;24(3):229-35. doi: 10.1123/jsr.2013-0114. Epub 2015 May 1. PMID 25933060
- [Background] Rogan S, Wust D, Schwitter T, Schmidtbleicher D. Static stretching of the hamstring muscle for injury prevention in football codes: a systematic review. Asian J Sports Med. 2013 Mar;4(1):1-9. Epub 2012 Nov 20. PMID 23785569
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777